CLINICAL TRIAL: NCT00463801
Title: A Multicentre, Open Label, Uncontrolled Clinical Trial to Evaluate Efficacy and Safety of Daptomycin for the Treatment of Complicated Skin and Skin-Structure Infections (cSSTI) Caused by Methicillin-resistant Staphylococcus Aureus (MRSA)
Brief Title: Safety and Efficacy of Daptomycin for the Treatment of Complicated Skin and Skin-structure Infections
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Because of inadequate accrual.
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCBC134AIT01
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Results first posted 2010-12-23 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Staphylococcal Skin Infections
Keywords: Complicated Skin and Skin-Structure Infections, Daptomycin, MRSA, Diabetic Foot, Abscess, Cellulitis; Complicated skin and skin-structure infections
MeSH Terms: conditions — Staphylococcal Skin Infections; Diabetic Foot; Abscess; Cellulitis | interventions — Daptomycin

ARMS (1):
- Daptomycin (Experimental): 350 mg of Daptomycin was supplied as sterile lyophilized powder in glass vials. Each vial was to be reconstituted with 7 mL of normal saline or water for injection, to give a 50 mg/mL drug concentration. Daptomycin was to be administered as a 30-minute intravenous infusion, once daily for at least 7 days, at the dose of 4 mg/Kg, up to a maximum of 14 days.
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Daptomycin

SUMMARY:
This study will evaluate the safety and efficacy of daptomycin against complicated skin and skin-structure infections in adults

ELIGIBILITY:
Inclusion criteria:

* Subjects with a diagnosis of complicated skin and skin-structure infections (cSSTI) defined as infection normally requiring surgical/local debridement of sufficient severity to warrant hospitalization and intravenous antimicrobial treatment
* Infection to be due to Gram-positive bacteria
* Hospitalized subjects
* Written informed consent
* Female patients of childbearing potential must have a negative pregnancy test urine or serum at baseline and must use effective contraception throughout the study period.

Exclusion criteria:

* Complicated skin and skin-structure infections of the following categories:
* Infected burns
* Severely impaired arterial blood supply
* Decubitus ulcers
* Infected diabetic foot ulcers associated with osteomyelitis
* Infected human or animal bites
* Perirectal abscess
* Necrotising fasciitis or gangrene
* Infections expected to require more than 14 days of intravenous antimicrobial therapy
* Skin and/or skin structure infection that can be treated by surgery alone
* Infections associated with a permanent prosthetic device that will not be removed within 2 days of study enrollment
* Uncomplicated skin or soft tissue infection
* Documented bacteremia at baseline
* Concomitant infection nearby the site of infection at baseline, potentially interfering with the evaluations
* Hospitalization for conditions related to rhabdomyolysis
* Human immunodeficiency virus (HIV) with cluster of differentiation (CD) < 200 or < 14%
* Immune function alterations
* Lack of sufficient purulent material for culture and Gram test
* Systemic or local antibiotic administration with known anti-Gram positive activity in the preceding 48 hours
* Complicated skin and soft tissue infections (cSSTI) known or believed to be related to fungal, parasitic or viral infection
* Pneumonia
* Local or systemic known or suspected allergy to daptomycin
* Creatinine clearance < 30 mL/min
* Severe liver damage (Child-Pugh class C) or Alanine transaminase (ALT) and/or Aspartate aminotransferase (AST) > 3 x Upper limit of normal (ULN) and/or bilirubin > 1.5 x ULN
* Use of any experimental drugs in the preceding 30 days
* Severe medical conditions that in the investigator's opinion could counter indicate participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-01; Primary Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (2):
- Italy (2):
  - Novartis Italy, Novartis Italy
  - Novartis Italy, Saronno

RESULTS

PARTICIPANT FLOW:
Groups:
- Daptomycin Intravenous: 350 mg of Daptomycin was supplied as sterile lyophilized powder in glass vials. Each vial was to be reconstituted with 7 mL of normal saline or water for injection, to give a 50 mg/mL drug concentration. Daptomycin was to be administered as a 30-minute intravenous infusion, once daily for at least 7 days, at the dose of 4 mg/Kg, up to a maximum of 14 days.
Period: Overall Study
Arm/Group | Daptomycin Intravenous
Started | 52
Completed | 39
Not Completed | 13
Not completed — Protocol Violation | 1
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 5
Not completed — No longer require therapy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Daptomycin Intravenous
Number analyzed (Participants) | 52
Age, Customized [Number; unit: participants]
  Age 27-88 years | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Clinical Success at the Day 7 (D7) and Day 14 (D14) Visit After Treatment Start
Description: Primary objective of the study was to evaluate the efficacy of intravenous (IV) daptomycin in the treatment of complicated skin and soft tissue infections (cSSTI) caused by methicillin-resistant Staphylococcus aureus (MRSA), as assessed by measuring the clinical success rate achieved at the day 7 and day 14 visit (D7, D14) after treatment start. Clinical success is defined as complete resolution of signs and symptoms of infection, or clinical improvement, i.e. partial resolution of signs and symptoms so that no further antibacterial treatment was required.
Time Frame: at Day 7 and 14
Population: Intention to treat (ITT) and safety population: all patients who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Daptomycin Intravenous
Number analyzed (Participants) | 52
Participants | 0

2. Secondary Outcome: Efficacy Assessed as Success After 4, 7, 10 and 14 Days of Treatment With Daptomycin on Infecting Gram Positive Bacteria
Description: To evaluate the microbiological efficacy of intravenous (IV) daptomycin in the treatment of complicated skin and soft tissue infections (cSSTI) caused by methicillin-resistant Staphylococcus aureus (MRSA), as assessed by measuring the proportion of patients achieving eradication of the Gram-positive baseline organisms at the study visits on D4, D7, D10, and D14. Microbiological success is documented eradication of baseline Gram-positive organism or presumed eradication defined as clinical success and no culture performed because of absence of drainage or other material for culture.
Time Frame: At day 4, 7, 10 and 14
Reporting Status: Not Posted

3. Secondary Outcome: Efficacy Assessed as Percentage of Patients With Clinical Success at Day 4 and 10
Description: To evaluate the efficacy of intravenous (IV) daptomycin in the treatment of complicated skin and soft tissue infections (cSSTI) caused by methicillin-resistant Staphylococcus aureus (MRSA), as assessed by measuring the clinical success rate achieved at the interim visits on day 4 (D4) and day 10 (D10) after treatment start. Clinical success is defined as complete resolution of signs and symptoms of infection, or clinical improvement, i.e. partial resolution of signs and symptoms so that no further antibacterial treatment was required.
Time Frame: At day 4 and 10
Reporting Status: Not Posted

4. Secondary Outcome: Efficacy Assessed by Duration of Treatment With Daptomycin Intravenous
Time Frame: At day 14
Reporting Status: Not Posted

5. Secondary Outcome: Efficacy Assessed by Time of Resolution of Infection
Description: Time to resolution of signs and symptoms of infection, time to resolution of fever (oral or tympanic temperature ≤37.5°C).
Time Frame: At day 14
Reporting Status: Not Posted

6. Secondary Outcome: Safety Assessed by Hematological and Biochemical Tests, Urinalysis, and Recording and Follow-up of Emerging AE and SAE
Time Frame: At day 14
Reporting Status: Not Posted

7. Secondary Outcome: Evaluated Resource Utilization and Calculated Overall Treatment Cost (Including Treatment Period and Follow-up Period)
Time Frame: at day 14 and follow up day i.e. day 30
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- All Patients: All patients
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 4/52
Other Adverse Events (participants affected / at risk) | 6/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=52)
Cellulitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=52)
Anaemia (Blood and lymphatic system disorders) | 3
Transaminases increased (Investigations) | 3

LIMITATIONS AND CAVEATS:
Inadequate accrual caused the premature study termination and the insufficient sample size, therefore none of the planned study analyses were performed; nor were any tabulations with descriptive statistics were provided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.